CLINICAL TRIAL: NCT07364526
Title: Non-invasive Preimplantation Genetic Screening (niPGTA) in Oocyte Donation Patients.
Brief Title: Non-Invasive Preimplantation Genetic Screening for Aneuploidies and Clinical Outcomes in Egg Donation Patients
Acronym: niPGTAdon
Status: Recruiting | Type: Observational
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Belen Lledo, Director, Instituto Bernabeu
Other Study IDs: IBB23
Record Dates: First submitted 2026-01-14; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: IVF
Keywords: niPGTA

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — spent medium
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preimplantation genetic testing for aneuploidies (PGT-A) is commonly used in IVF but requires embryo biopsy and shows limited benefit in egg donation cycles. Non-invasive PGT-A (niPGTA), based on the analysis of cell-free embryonic DNA in spent culture media, offers a promising biopsy-free alternative. This prospective, blinded study in egg donation cycles will evaluate whether niPGTA-detected aneuploidy is associated with implantation failure and pregnancy loss, assessing its potential clinical value as a non-invasive embryo selection tool.

DETAILED DESCRIPTION:
Preimplantation genetic testing for aneuploidies (PGT-A) is widely used in IVF to improve embryo selection and pregnancy outcomes. However, it requires invasive embryo biopsy and has not shown clear benefit in egg donation cycles, where embryos originate from young donors with lower aneuploidy rates. Non-invasive PGT-A (niPGTA), based on the analysis of cell-free embryonic DNA released into the culture medium, represents a promising alternative that avoids embryo biopsy.

This prospective, blinded, non-selection study will include women undergoing egg donation treatment. Embryos will be selected for transfer using standard morphological criteria only, while niPGTA results will not influence clinical decisions. After embryo transfer, the spent culture medium will be collected and analyzed using next-generation sequencing to determine the presence of chromosomal aneuploidies.

The study aims to evaluate whether aneuploidy detected by niPGTA is associated with implantation failure, biochemical pregnancy loss, and clinical miscarriage. By comparing niPGTA results between embryos that result in pregnancy and those that do not, this project will assess the potential clinical value of niPGTA as a non-invasive embryo selection tool in egg donation cycles.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 50 years old who are oocyte recipients.
* Signed consent form
* Transfer of a single blastocyst-stage embryo
* Male with normal sperm FISH

Exclusion Criteria:

* Uterine malformations
* Abnormal karyotypes in either partner
* Failure to sign informed consent

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Recipient of embryo transfer
Study Population: Patients who are going to undergo an oocyte donation cycle, who meet the inclusion/exclusion criteria and who sign the informed consent form
Sampling Method: Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2026-02-26 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | 9 months from enrolment

SECONDARY OUTCOMES:
Pregnancy rate | 2 weeks from enrolment
Miscarriage rate | 12 weeks from enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Bernabeu, Alicante, Spain